CLINICAL TRIAL: NCT06097039
Title: Fetuin-A, a Promising Serum Biomarker for Diagnosis of Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Fetuin-A, a Promising Serum Biomarker for Diagnosis of Non-Alcoholic Fatty Liver Disease
Acronym: NAFLD
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Collaborators: Suez University (Other); Benha University (Other)
Responsible Party: Sponsor
Other Study IDs: Diagnosis of the NAFLD
Record Dates: First submitted 2023-09-24; First posted 2023-10-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: fetuin-A; fibroscan; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NAFLD subjects group: The group including 50 cases with NAFLD, the diagnosis was based on abdominal U/S and Fibroscan with CAP with or without elevated liver enzymes
  Interventions: Device: abdominal U/S; Device: Fibroscan with Controlled Attenuated Parameter (CAP scan):
- Healthy subjects group: The group including 50 healthy subjects as a control group with normal liver in transabdominal ultrasonography and normal liver enzymes
  Interventions: Device: abdominal U/S; Device: Fibroscan with Controlled Attenuated Parameter (CAP scan):

INTERVENTIONS:
Device: abdominal U/S — A convex transducer with a frequency range of 2-5 MHz was used for ultrasound. Based on a visual study of the intensity of the echogenicity and under the assumption that the gain setting is optimal, various (0-3) degrees of steatosis have been proposed. Grade I occurs when the echogenicity is simply increased; grade II occurs when the echogenic liver obscures the echogenic walls of the portal vein branches; and grade III occurs when the echogenic liver obscures the diaphragmatic contour.
Device: Fibroscan with Controlled Attenuated Parameter (CAP scan): — Using FibroScan502 (Echosens, Paris, France), liver stiffness measurement (LSM) and CAP were acquired. Before the treatment, all subjects will be instructed to fast for at least 8 hours.
  The median of 10 measurements served as the LSM score, which was only deemed credible if at least 10 successful acquisitions were made and the IQR-to-median ratio of the 10 acquisitions was below 30%. If 10 successful acquisitions are made, CAP measures were deemed trustworthy and taken into account in the final analysis.
  CAP graded the degree of hepatic steatosis using the M probe in accordance with standard cut-off values (S1=222-232; S2= 233-289; and S3 290 dB/m).

SUMMARY:
The work investigate the role of fetuin-A in the diagnosis and assessment of the severity of non-alcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
The prevalence of nonalcoholic fatty liver disease (NAFLD), which has recently become one of the most prevalent chronic liver illnesses, is about 25% worldwide. NAFLD is a progressive liver disease that can cause fibrosis and ultimately cirrhosis, in contrast to simple hepatic steatosis, which is considered to be a benign condition. The sole way to diagnose NAFLD and stage liver fibrosis has historically been a liver biopsy. There are a number of issues with this method, though. A liver biopsy is a painful and invasive diagnostic procedure that carries a risk of consequences.

Fetuin-A, also called the 2-Heremans-Schmid glycoprotein, belongs to the fetuin group of serum-binding proteins and is largely produced by hepatocytes. It is a phosphorylated glycoprotein. Fetuin-A can cause insulin resistance in the target organs, including the liver and skeletal muscle, as it is an endogenous tyrosine kinase inhibitor. A strong correlation between the level of circulating fetuin-A and the onset and progression of NAFLD has been described by accumulating lines of evidence, but the findings have been contradictory.

The investigators want to find out how fetuin-A affects the diagnosis and evaluation of the severity of non-alcoholic fatty liver disease (NAFLD) and to reveal the relationship between fetuin-A and the NAFLD fibrosis score (NFS).

ELIGIBILITY:
Inclusion Criteria:

* patients who were admitted to the university hospitals with inclusion criteria

Exclusion Criteria:

* Patients who are younger than 18 years old,
* Patients with a history of high alcohol consumption (more than 40 g/day for men and 20 g/day for women) over the previous five years,
* Patients who have concurrent hepatitis B and hepatitis C viral infections
* Patients with hepatobiliary malignancy, Wilson's disease, alpha-one antitrypsin deficiency, and autoimmune hepatitis,
* Pregnant women
* Patients who take steatogenic pharmaceuticals including amiodarone, valproic acid, antiretrovirals, methotrexate, and tetracyclines, or NAFLD treatments like vitamin E, metformin, and thiazolidinediones

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who were admitted to the university hospitals with inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
To assess fetuin-A serum concentration | 30 minutes.
  Serum fetuin-A serum concentrations of fetuin-A was measured by using a human fetuin-A sandwich enzyme-linked immunosorbent assay (ELISA) kit.
To measure liver stiffness and fibrosis degree | 30 minutes
  liver stiffness measurement (LSM) and fibrosis degreewere obtained using FibroScan502 (Echosens, Paris, France). The LSM score was represented by the median of 10 measurements and was considered reliable only if at least 10 successful acquisitions were obtained and the IQR-to-median ratio of the 10 acquisitions was ≤30%.
Number of participants with fetuin-A serum concentration and liver stiffness degree using FibroScan | 30 minutes
  Number of participants with fetuin-A serum concentration and liver stiffness degree using FibroScan

CONTACTS AND LOCATIONS:
Overall Officials: Amira A Othman, PhD, Principal Investigator — Lecturer of Internal Medicine
Locations (1):
- Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No
to keep participant privacy

REFERENCES:
- [Background] Friedman SL, Neuschwander-Tetri BA, Rinella M, Sanyal AJ. Mechanisms of NAFLD development and therapeutic strategies. Nat Med. 2018 Jul;24(7):908-922. doi: 10.1038/s41591-018-0104-9. Epub 2018 Jul 2. PMID 29967350
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Result] WHO Expert Consultation. Appropriate body-mass index for Asian populations and its implications for policy and intervention strategies. Lancet. 2004 Jan 10;363(9403):157-63. doi: 10.1016/S0140-6736(03)15268-3. PMID 14726171
- [Result] Sasso M, Tengher-Barna I, Ziol M, Miette V, Fournier C, Sandrin L, Poupon R, Cardoso AC, Marcellin P, Douvin C, de Ledinghen V, Trinchet JC, Beaugrand M. Novel controlled attenuation parameter for noninvasive assessment of steatosis using Fibroscan((R)): validation in chronic hepatitis C. J Viral Hepat. 2012 Apr;19(4):244-53. doi: 10.1111/j.1365-2893.2011.01534.x. Epub 2011 Oct 13. PMID 22404722
- [Result] Schwimmer JB, Middleton MS, Behling C, Newton KP, Awai HI, Paiz MN, Lam J, Hooker JC, Hamilton G, Fontanesi J, Sirlin CB. Magnetic resonance imaging and liver histology as biomarkers of hepatic steatosis in children with nonalcoholic fatty liver disease. Hepatology. 2015 Jun;61(6):1887-95. doi: 10.1002/hep.27666. Epub 2015 Feb 5. PMID 25529941
- [Derived] Elhoseeny MM, Abdulaziz BA, Mohamed MA, Elsharaby RM, Rashad GM, Othman AAA. Fetuin-A: a relevant novel serum biomarker for non-invasive diagnosis of metabolic dysfunction-associated steatotic liver disease (MASLD): a retrospective case-control study. BMC Gastroenterol. 2024 Jul 18;24(1):226. doi: 10.1186/s12876-024-03310-y. PMID 39026172